CLINICAL TRIAL: NCT07325240
Title: 24-hour Effect Of Rocklatan Compared With Latanoprost In Open Angle Glaucoma And Ocular Hypertension Patients
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Arthur J. Sit, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-012250
Record Dates: First submitted 2026-01-01; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — netarsudil; Latanoprost; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- netarsudil-latanoprost arm (Experimental)
  Interventions: Drug: Netarsudil 0.01%/latanoprost 0.005% ophthalmic solution
- latanoprost arm (Active Comparator)
  Interventions: Drug: Latanoprost 0.005% Ophthalmic Solution

INTERVENTIONS:
Drug: Netarsudil 0.01%/latanoprost 0.005% ophthalmic solution — Subjects will receive netarsudil-latanoprost fixed combination ophthalmic solution 0.02%/0.005% in one eye and compare it to latanoprost 0.005% in the contralateral eye
  Arms: netarsudil-latanoprost arm
Drug: Latanoprost 0.005% Ophthalmic Solution — latanoprost 0.005% solution will be applied in the contralateral eye, once daily, QD (PM) for 14 days
  Arms: latanoprost arm

SUMMARY:
The purpose of this study is to evaluate the effect on 24-hour IOP reduction of netarsudil-latanoprost fixed combination in one eye compared to latanoprost alone in the contralateral eye, dosed daily, 1 drop at night (QD, PM) in adult subjects, at least 18 years of age, with open angle glaucoma (OAG) or ocular hypertension (OHT).

DETAILED DESCRIPTION:
This will be a double-masked, paired-contralateral, descriptive study to evaluate the effect on 24-hour IOP reduction of netarsudil-latanoprost fixed combination in one eye compared to latanoprost alone in the contralateral eye, dosed daily, 1 drop at night (QD, PM) in adult subjects, at least 18 years of age, with open angle glaucoma (OAG) or ocular hypertension (OHT). Study medication will be administered for 14 consecutive days, although the total time of subject participation in the study (including washout from prior treatment, if necessary) may be up to 10 weeks.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of OHT or mild-to-moderate OAG in both eyes (OAG in one eye and OHT in the fellow eye is acceptable) based on VF, OCT and dilated fundus examination within one year of the screening visit.
* Both eyes must qualify for the study with an IOP of ≥18 mmHg but ≤34 mmHg on history or at the screening visit
* Be able and willing to provide signed informed consent and follow study instructions
* Ability to cooperate with the examinations required for the study and be able to attend all study visits
* If a contact lens wearer, willing to remove contact lenses at least 24 hours prior to each of the study visits.
* Best-corrected visual acuity (BCVA) using ETDRS chart of +0.4 logMAR units (Snellen equivalent ~ 20/50) or better in each eye

Exclusion Criteria

Ocular:

* Subjects with narrow angles (3 quadrants with Grade 2 or less according to Shaffer Scale), angle closure or a history of angle closure, or peripheral iridotomy in either eye
* Severe glaucomatous damage
* Difference in IOP between eyes > 4 mmHg (unmedicated) at any baseline time point
* Use of more than two ocular hypotensive medications within 30 days of screening
* Chronic or recurrent inflammatory eye diseases in either eye
* Ocular infection or ocular inflammation in the past 3 months in either eye
* Ocular trauma other than corneal abrasion within the past 6 months in either eye
* Clinically significant retinal disease (e.g., severe diabetic retinopathy, exudative or severe non-exudative macular degeneration, macular edema, retinal vein or artery occlusion) in either eye
* Cornea pathologic changes preventing reliable measurement (e.g., scarring, opacity, edema, keratoconus) in either eye
* Myopia greater than -6.00D, or hyperopia greater than +2.00D in either eye
* Central corneal thickness less than 480 μm or greater than 620 μm in either eye
* Previous intraocular surgery other than routine uncomplicated cataract surgery in either eye
* Previous glaucoma intraocular surgery or glaucoma laser procedures (except SLT performed more than 6 months ago) in either eye
* Unilateral intraocular surgery or glaucoma laser procedures
* Previous corneal refractive surgery in either eye (eg, radial keratotomy, PRK, LASIK, corneal cross-linking, etc.)
* Severe dry eye in either eye
* Use of ocular medications in either eye within 30 days of screening, with the exception of IOP-lowering medications (which must be washed out according to the provided schedule), and lubricating drops for dry eye (which may be used throughout the study)
* Known hypersensitivity to any component of the formulation (eg, benzalkonium chloride, etc.), or to topical anesthetic

Systemic:

* Clinically significant systemic diseases which might interfere with the study
* Participation in any interventional study within 30 days prior to screening visit
* Changes of systemic medication that could have an effect on IOP within 30 days prior to screening, or anticipated during the study including, β-adrenergic antagonists, α-adrenergic agonists and antagonists, angiotensin converting enzyme (ACE) inhibitors, angiotensin II receptor blockers
* Recent change in medications that are known to affect IOP within 30 days prior to the screening visit and during the study including: systemic/inhaled steroids, calcium channel blockers, diuretics, and vasodilators
* Women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control. An adult woman is considered to be of childbearing potential unless she is one year post-menopausal or three months post-surgical sterilization. All females of childbearing potential must have a negative pregnancy test result at the screening examination and must not intend to become pregnant during the study
* Subjects with a known hypersensitivity or contraindications to any of the ingredients in the study medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change in mean Intraocular Pressure (IOP) | Change in mean IOP after 2 weeks of treatment with Latanoprost compared to baseline
  Change in mean IOP from baseline at each time point for Latanoprost
Change in mean IOP | Change in mean IOP after 2 weeks of treatment with Rocklatan compared to baseline
  Change in mean IOP from baseline at each time point for Rocklatan
Change in mean IOP | Change in mean IOP from baseline after 2 weeks of treatment with latanoprost minus change in mean IOP from baseline after 2 weeks of treatment with Rocklatan
  Change in mean IOP from Latanoprost at each time point for Rocklatan

SECONDARY OUTCOMES:
Change in mean nocturnal IOP | Mean nocturnal IOP will be calculated based on the time points during the sleeping hours (11 PM - 7 AM) after 2 weeks of treatment with Latanoprost compared to baseline
  Change in mean nocturnal IOP (both absolute and % change) from baseline for Latanoprost
Change in mean nocturnal IOP | Mean nocturnal IOP will be calculated based on the time points during the sleeping hours (11 PM - 7 AM) after 2 weeks of treatment with Rocklatan compared to baseline
  Change in mean nocturnal IOP (both absolute and % change) from baseline for Rocklatan
Change in mean diurnal IOP | Mean diurnal IOP will be calculated based on the time points during the sleeping hours (7 AM - 11 PM) after 2 weeks of treatment with Latanoprost compared to baseline
  Change in mean diurnal IOP (both absolute and % change) from baseline for Latanoprost
Change in mean diurnal IOP | Mean diurnal IOP will be calculated based on the time points during the sleeping hours (7 AM - 11 PM) after 2 weeks of treatment with Rocklatan compared to baseline
  Change in mean diurnal IOP (both absolute and % change) from baseline for Rocklatan

OTHER OUTCOMES:
24-hour IOP variability | During the time period of analysis, approximately 18 months
  24-hour IOP variability based on standard deviation and range of measurements from 12 time points over a 24-hour period, and circadian amplitude from cosinor analysis of the 24-hour curve
Diurnal IOP variability | During the time period of analysis, approximately 18 months
  Diurnal IOP variability based on standard deviation and range of measurements during the waking period
Nocturnal IOP variability | During the time period of analysis, approximately 18 months
  Nocturnal IOP variability based on standard deviation and range of measurements during the sleeping period

CONTACTS AND LOCATIONS:
Overall Officials: Arthur J Sit, MD, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nelson W, Tong YL, Lee JK, Halberg F. Methods for cosinor-rhythmometry. Chronobiologia. 1979 Oct-Dec;6(4):305-23. No abstract available. PMID 548245
- [Background] Asrani S, Bacharach J, Holland E, McKee H, Sheng H, Lewis RA, Kopczynski CC, Heah T. Fixed-Dose Combination of Netarsudil and Latanoprost in Ocular Hypertension and Open-Angle Glaucoma: Pooled Efficacy/Safety Analysis of Phase 3 MERCURY-1 and -2. Adv Ther. 2020 Apr;37(4):1620-1631. doi: 10.1007/s12325-020-01277-2. Epub 2020 Mar 12. PMID 32166538
- [Background] Brubaker JW, Teymoorian S, Lewis RA, Usner D, McKee HJ, Ramirez N, Kopczynski CC, Heah T. One Year of Netarsudil and Latanoprost Fixed-Dose Combination for Elevated Intraocular Pressure: Phase 3, Randomized MERCURY-1 Study. Ophthalmol Glaucoma. 2020 Sep-Oct;3(5):327-338. doi: 10.1016/j.ogla.2020.05.008. Epub 2020 Jun 4. PMID 32768361
- [Background] Peace JH, McKee HJ, Kopczynski CC. A Randomized, Phase 2 Study of 24-h Efficacy and Tolerability of Netarsudil in Ocular Hypertension and Open-Angle Glaucoma. Ophthalmol Ther. 2021 Mar;10(1):89-100. doi: 10.1007/s40123-020-00322-1. Epub 2020 Nov 26. PMID 33244711
- [Background] Sit AJ, Nau CB, McLaren JW, Johnson DH, Hodge D. Circadian variation of aqueous dynamics in young healthy adults. Invest Ophthalmol Vis Sci. 2008 Apr;49(4):1473-9. doi: 10.1167/iovs.07-1139. PMID 18385065
- [Background] Nau CB, Malihi M, McLaren JW, Hodge DO, Sit AJ. Circadian variation of aqueous humor dynamics in older healthy adults. Invest Ophthalmol Vis Sci. 2013 Nov 15;54(12):7623-9. doi: 10.1167/iovs.12-12690. PMID 24243986
- [Background] Sit AJ, Weinreb RN, Crowston JG, Kripke DF, Liu JH. Sustained effect of travoprost on diurnal and nocturnal intraocular pressure. Am J Ophthalmol. 2006 Jun;141(6):1131-3. doi: 10.1016/j.ajo.2006.01.049. PMID 16765686
- [Background] Brubaker RF. Flow of aqueous humor in humans [The Friedenwald Lecture]. Invest Ophthalmol Vis Sci. 1991 Dec;32(13):3145-66. PMID 1748546
- [Background] Tung JD, Tafreshi A, Weinreb RN, Slight JR, Medeiros FA, Liu JH. Twenty-four-hour effects of bimatoprost 0.01% monotherapy on intraocular pressure and ocular perfusion pressure. BMJ Open. 2012 Aug 23;2(4):e001106. doi: 10.1136/bmjopen-2012-001106. Print 2012. PMID 22918671
- [Background] Liu JH, Medeiros FA, Slight JR, Weinreb RN. Diurnal and nocturnal effects of brimonidine monotherapy on intraocular pressure. Ophthalmology. 2010 Nov;117(11):2075-9. doi: 10.1016/j.ophtha.2010.03.026. Epub 2010 Jul 21. PMID 20663566
- [Background] Liu JH, Medeiros FA, Slight JR, Weinreb RN. Comparing diurnal and nocturnal effects of brinzolamide and timolol on intraocular pressure in patients receiving latanoprost monotherapy. Ophthalmology. 2009 Mar;116(3):449-54. doi: 10.1016/j.ophtha.2008.09.054. Epub 2009 Jan 20. PMID 19157559
- [Background] Liu JH, Kripke DF, Weinreb RN. Comparison of the nocturnal effects of once-daily timolol and latanoprost on intraocular pressure. Am J Ophthalmol. 2004 Sep;138(3):389-95. doi: 10.1016/j.ajo.2004.04.022. PMID 15364220
- [Background] Sit AJ, Gupta D, Kazemi A, McKee H, Challa P, Liu KC, Lopez J, Kopczynski C, Heah T. Netarsudil Improves Trabecular Outflow Facility in Patients with Primary Open Angle Glaucoma or Ocular Hypertension: A Phase 2 Study. Am J Ophthalmol. 2021 Jun;226:262-269. doi: 10.1016/j.ajo.2021.01.019. Epub 2021 Jan 29. PMID 33524367
- [Background] Kazemi A, McLaren JW, Kopczynski CC, Heah TG, Novack GD, Sit AJ. The Effects of Netarsudil Ophthalmic Solution on Aqueous Humor Dynamics in a Randomized Study in Humans. J Ocul Pharmacol Ther. 2018 Jun;34(5):380-386. doi: 10.1089/jop.2017.0138. Epub 2018 Feb 22. PMID 29469601
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials